CLINICAL TRIAL: NCT03597971
Title: A Phase I, Randomized, Double Blind, Placebo-controlled, Dose-escalating Study of the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of HMPL004-6599 in Healthy Male Volunteers
Brief Title: HMPL004-6599 Phase I Dose-escalating Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nutrition Science Partners Limited (Industry)
Collaborators: Hutchison Medipharma Limited (Industry); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-599-00AU1
Record Dates: First submitted 2018-05-03; First posted 2018-07-24 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo-controlled, dose-escalating, single dose study in healthy volunteers followed by a double blind, randomized, placebo-controlled, dose-escalating, multiple dose study in healthy volunteers.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: experimental (Experimental): Subjects will receive HMPL004-6599 or matching placebo on Day 1. This will be administered under fed conditions with a standard meal, according to the randomization schedule. Dose levels may be repeated, or reduced if deemed appropriate by the Safety Monitoring Committee (SMC).
  Interventions: Drug: HMPL004-6599
- Part A: placebo (Placebo Comparator): Subjects will receive matching placebo on Day 1. This will be administered under fed conditions with a standard meal, according to the randomization schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMPL004-6599 — For each cohort, 6 subjects will receive HMPL004-6599
  Arms: Part A: experimental
Drug: Placebo — For each cohort, 2 subjects will receive placebo
  Arms: Part A: placebo

SUMMARY:
To assess the safety and tolerability of single and multiple doses of HMPL004-6599 in healthy male volunteers

DETAILED DESCRIPTION:
This is a Phase I study with two parts:

Part A: Double blind, randomized, placebo-controlled, dose-escalating, single dose study in healthy volunteers.

Subjects will receive a single dose of up to 1800 mg HMPL004-6599 or matching placebo on Day 1. The planned dose levels are: 600, 1200, and 1800 mg under fed conditions with a standard meal, according to the randomization schedule. Dose levels may be repeated, or reduced if deemed appropriate by the Safety Monitoring Committee (SMC).

Part B: Double blind, randomized, placebo-controlled, dose-escalating, multiple dose study in healthy male volunteers.

Dose levels in Part B for 14 days are planned as 200mg TID, 400mg TID, 600mg BID and 600mg TID. These dose were jointly decided by the PI, SMC and the Sponsor based on the results from Part A. On day 14, only one dose in the morning will be administrated for all cohorts. Dose levels may be repeated, or reduced if deemed appropriate by the Safety Monitoring Committee (SMC).

In Part A, cohort 1 will consist of a blinded sentinel group of two subjects; one subject will receive HMPL004-6599 and the other will receive placebo, at least 24 hours prior to dosing the remaining 6 subjects in the cohort. The remaining subjects will only be dosed after review of available safety data from the sentinel subjects.

During Part A and Part B, PK sample collections will take place. During Part A, a full PK profile will be measured throughout Day 1. Samples will be collected from pre-dose to 24 hours post dose.

Part B PK sample collection is based on Part A study data. A full PK testing of plasma samples from pre-dose to 8 (TID) or 12 (BID) hours post dose will be collected on the first and last dosing days. Stool samples produced at baseline before dose and day 14-15 post last dose will be collected.

Concentrations of Andrographolide (AND), 14-deoxy-11,12- didehydroandrographolide (DDAND), HM5013620, neoandrographolide (NAND) and 14-deoxyandrographolide (DAND) in plasma (Part A and B) and fecal samples (Part B) will be determined for each dose level.

The plasma samples will be analyzed at the lab contracted by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following for inclusion in the trial:

1. Informed consent must be obtained in writing for all subjects before enrollment into the study.
2. Healthy male subjects aged 18 to 45 years inclusive at the time of screening.
3. Body mass index ≥19.0 and ≤ 30.0 kg/m2
4. No clinically significant abnormalities as determined by medical history and physical examination, especially with regard to the liver, bile and gastrointestinal systems.
5. No clinically significant laboratory values and urinalysis, as determined by the Clinical Investigator.
6. No clinically significant findings in ECG, blood pressure and heart rate, as determined by the Clinical Investigator.
7. Willing to comply with the contraceptive requirements of the study and must not donate sperm during the study and for 3 months afterwards. Subjects must agree to use a condom or to abstain from sexual intercourse throughout the trial and for 3 months afterwards.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Family history of premature Coronary Heart Disease
2. History of immunosuppression or opportunistic infections or receipt of a live virus vaccination within the 3 months prior to screening.
3. Subjects at risk for tuberculosis (TB), specifically subjects with:

   1. Clinical or laboratory evidence of active TB
   2. History of active TB unless there is documentation that the prior anti-TB treatment was appropriate in duration and type
   3. Latent TB which has not been successfully treated
4. History of hypertension requiring treatment.
5. Any condition requiring the regular use of any medication.
6. Exposure to prescription medications within 30 days prior to Day 1.
7. Exposure to any other medication, including over-the counter medications, herbal remedies and vitamins 14 days prior to first dose (except for paracetamol).
8. Participation in another study with any investigational drug in the 30 days preceding Day 1 of the study or in the exclusion period of any previous study with investigational drugs.
9. Treatment in the previous 3 months with any drug known to have a well-defined potential for toxicity to a major organ. Once-off medication such as paracetamol or any medication deemed not clinically significant by the principal investigator can be permitted.
10. Current smoker of more than 10 cigarettes or equivalent / day during past 3 months prior to commencing the study and unable to completely stop smoking during the study.
11. Symptoms of a clinically significant illness in the 3 months before the study.
12. Presence or sequelae of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
13. Chronic constipation or diarrhea, irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), Hemorrhoids or anal diseases with regular or recent presence of blood in feces.
14. History of significant allergic disease (e.g. Allergic to medications) and acute phase of allergic rhinitis in the previous 2 weeks before randomization/enrollment or any food allergy.
15. Blood or plasma donation of no more than 470 ml during the past 30 days (equivalent to the standard blood donation in Australia) before randomization/enrollment and/or more than 50 ml in the 2 weeks prior to screening.
16. Known positive test for human immunodeficiency virus (HIV).
17. Known positive test for hepatitis B or C, unless caused by immunization.
18. Current evidence of drug abuse or history of drug abuse within one year before randomization/enrollment.
19. History of alcohol abuse or active alcoholism with average weekly alcohol intake that exceeds 21 units.
20. Mental condition rendering the subject incapable to understand the nature, scope, and possible consequences of the study.
21. Adults under guardianship and people with restriction of freedom by administrative or legal decisions.
22. Unlikely to comply with the clinical study protocol; e.g. uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study.
23. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
24. Known allergy to plants of the Acanthaceae family.
25. Those Subjects who are Vegetarian due to the requirements of the Standard Meal.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects aged 18 to 45 years of age inclusive at the time of screening.
Enrollment: 32 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Part A: single dose; Part B: 21 days
  A primary objective of this study is to assess the safety of a single dose of up to 1800 mg in Part A (evaluated in planned steps of 600, 1200, and 1800 mg HMPL004-6599 under fed conditions of a standard meal), followed by multiple doses of up to 1800mg in Part B (evaluated in planned steps of 200mg TID, 400mg TID, 600mg BID and 600mg TID HMPL004-599 under fed conditions of a standard meal for 14 days ) in healthy male volunteers.
  The occurrence of Serious Adverse Events and Adverse Events will be evaluated during the study in order to determine this primary objective.
Incidence of Participants with Abnormal Laboratory Values | Part A: single dose; Part B: 21 days
  A further primary objective of this study is to assess the tolerability of a single dose of up to 1800 mg in Part A (evaluated in planned steps of 600, 1200, and 1800 mg HMPL004-6599 under fed conditions of a standard meal), followed by multiple doses of up to 1800mg in Part B (evaluated in planned steps of 200mg TID, 400mg TID, 600mg BID and 600mg TID HMPL004-599 under fed conditions of a standard meal for 14 days ) in healthy male volunteers.
  The occurrence of abnormal laboratory values will be reviewed during the study in order to determine this primary objective.

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Part A: single dose; Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the Cmax determination after single (Part A) and multiple (Part B) oral doses in healthy male volunteers.
Area Under The Concentration Time Curve Up To The Time 't' [AUC0-t] | Part A: single dose; Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the AUC0-t determination after single (Part A) and multiple (Part B) oral doses in healthy male volunteers.
Time of Maximum Plasma Drug Concentration [Tmax] | Part A: single dose; Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the Tmax determination after single (Part A) and multiple (Part B) oral doses in healthy male volunteers.
Area Under The Concentration Time Curve Up To The Last Data Point Above LOQ [AUClast] | Part A: single dose; Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the AUClast determination after single (Part A) and multiple (Part B) oral doses in healthy male volunteers.
Apparent Half-Life For Designated Elimination Phases [t1/2] | Part A: single dose; Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the t1/2 determination after single (Part A) and multiple (Part B) oral doses in healthy male volunteers.
Area Under The Concentration-Time Curve During Once Dosing Interval [AUCTau or AUC0-_] | Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the AUCTau or AUC0-_determination after multiple (Part B) oral doses in healthy male volunteers.
Minimum Observed Concentration [Cmin] | Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the AUCTau or AUC0-_determination after multiple (Part B) oral doses in healthy male volunteers.
Average Concentration [Cavg] | Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the Cavg determination after multiple (Part B) oral doses in healthy male volunteers.
%_Fluctuation | Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the %_Fluctuation determination after multiple (Part B) oral doses in healthy male volunteers.
Accumulation Ratio_obs | Part B: 21 days
  Plasma concentration of HMPL004-6599 to evaluate protocol specified Pharmacokinetic parameters. Where these PK parameters are derived from plasma concentrations of AND, DDAND, HM5013620, DAND and NAND and include but are not limited to the Accumulation Ratio_obs determination after multiple (Part B) oral doses in healthy male volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yan, MD, Study Director — Hutchison Medipharma Limited
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia